CLINICAL TRIAL: NCT01829555
Title: A Pilot Study Examining a Reinforcement Approach to Improve Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Yale University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-043-2; 1DP3DK097705 (NIH)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- contingency management (Experimental): The intervention will provide escalating financial reinforcement for self-monitored blood glucose testing.
  Interventions: Behavioral: contingency management

INTERVENTIONS:
Behavioral: contingency management — Participants will receive a voucher for each self-monitored blood glucose test completed during the target testing window, and a bonus amount for each day that 4 tests fall within the testing windows and are separated by more than 2 hours.

SUMMARY:
Glucose control is necessary to avoid the immediate and long-term adverse effects associated with type 1 diabetes, and frequent self-monitoring of blood glucose is the first important step to achieving glucose control. Data suggest that large proportions of adolescents and young adults fail to adhere to standard guidelines of self-monitored of blood glucose testing and have hemoglobin A1c levels >7.5%. A finite period of poor metabolic control can lead to increased risk of medical complications over an individual's lifespan, necessitating novel interventions to improve self-monitored blood glucose testing and metabolic control in emerging adults with type 1 diabetes. The investigators treatment approach, which provides direct tangible reinforcement for objective evidence of behavior change, is efficacious in decreasing substance use, reducing weight, and improving medication adherence.

The purpose of this project is to develop and pilot test an intervention based on behavioral economic principles for improving self-monitored blood glucose testing in young persons with type 1 diabetes. In this pilot study, patients will text in, via cell phones, each time they test, and a return text will inform them of reinforcer vouchers earned. The investigators will collect data on self-monitored blood glucose testing frequency and A1c levels preceding treatment initiation and throughout a 6 month treatment period. If promising, a randomized trial will lead to larger scale evaluations of reinforcement interventions alone, or in combination with multimodal treatment approaches, and it may be applied to other clinical issues such as adherence to continuous glucose monitoring. Importantly, this intervention can be administered remotely and in an automated fashion, allowing for widespread adoption if efficacious.

ELIGIBILITY:
Inclusion Criteria:

* age 15-21 years old
* diagnosis of type 1 diabetes (T1D) >12 months via ADA guidelines (Silverstein et al., 2005)
* average A1c >7.5% and <11% during the year before study entry, and most recent A1c >7.5% but <11%
* SMBG user with clinical recommendations to test >4 times/day
* past month SMBG <4 times/ day on average
* English speaking and able to read at >5th grade level

Exclusion Criteria:

* have a major psychiatric or neurocognitive disorder that would inhibit participation
* have a major visual impairment
* meet DSM-IV criteria for pathological gambling
* have a significant other medical condition that impacts diabetes management
* plan to switch insulin delivery mode (injection to pump or vice versa) in the next 12 months, or have recently switched
* are pregnant or trying to become pregnant
* are participating in another clinical trial

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change from baseline in number of self-monitoring of blood glucose tests conducted | 6 months

SECONDARY OUTCOMES:
change from baseline in hemoglobin A1c levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health; William Tamborlane, M.D., Principal Investigator — Yale University
Locations (1):
- Pediatric Endocrinology, Yale University, New Haven, Connecticut, United States